CLINICAL TRIAL: NCT02998086
Title: A Pilot Randomized Controlled Trial of the Promoting Resilience in Stress Management (PRISM) Intervention for Parents of Children With Cancer
Brief Title: PRISM for Parents of Children With Cancer Promoting Resilience in Stress Management (PRISM) Intervention for Parents of Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Abby Rosenberg, Associate Professor, Pediatrics, University of Washington, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SC-N120
Record Dates: First submitted 2016-12-13; First posted 2016-12-20 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Individual (1:1) (Experimental): Individual, 1:1 version of the Promoting Resilience in Stress Management for Parents (PRISM-P) intervention
  Interventions: Behavioral: Promoting Resilience in Stress Management
- Group (Experimental): Group-based version of the Promoting Resilience in Stress Management for Parents (PRISM-P) intervention
  Interventions: Behavioral: Promoting Resilience in Stress Management
- Usual Care (No Intervention): Usual non-directed psychosocial supportive care

INTERVENTIONS:
Behavioral: Promoting Resilience in Stress Management — Skills-based intervention designed to promote resilience resources
  Other Names: PRISM
  Arms: Group; Individual (1:1)

SUMMARY:
Parenting a child with cancer is highly stressful. The investigators have designed a promising parent-centered intervention to bolster parent resilience and reduce stress and distress. This study will test 2 formats of the intervention (individual or group-based) and compare them to usual care.

DETAILED DESCRIPTION:
Parenting a child with cancer is highly distressing. Both during and after cancer therapy, parents may suffer from poor mental health, risky health behaviors, and financial hardship, all of which may impact patients, siblings, and the family unit. Positive psychological resources can mitigate negative outcomes. In this regard, resilience is particularly important, describing an individual's ability to maintain psychological and/or physical well-being in the face of stress.

The investigators have previously described the "Promoting Resilience in Stress Management" (PRISM) intervention for adolescent and young adult patients with cancer. This brief, 1:1 intervention targets four "resilience resources" over approximately 3 months: skills in stress-management/mindfulness, goal-setting, cognitive restructuring, and meaning-making. Notably, every parent whose child received the PRISM requested a similar intervention for him- or herself. Hence, the investigators adapted two versions of the intervention for parents (the "PRISM-P"). First, using the same 1:1 format, they piloted the PRISM-P amongst 12 parents of children with cancer. Feedback was highly positive; however, many parents requested additional group-based social support. Second, they conducted a half-day symposium and administered small-group adaptations of the PRISM-P to 70 parents of children with serious illness. Feedback was again positive; however, the opportunity to develop individual skills was limited.

This application proposes a pilot Randomized Clinical Trial (RCT) to evaluate and compare these 2 formats of the PRISM-P with usual care, in order to determine optimal methodologies and preferences for future, larger studies. Consecutive eligible parents of children with newly diagnosed cancer will be randomly assigned to one of the 3 options (N=75 total, n=25 per arm). Secondary aims will assess parent-reported stress, burden of care, hope, goals, optimism, benefit-finding, psychological distress, and health behaviors, and ongoing perceptions of usefulness, feasibility, and preference.

ELIGIBILITY:
Inclusion Criteria: Parents of children who:

* Are aged 2-24 years
* Have been diagnosed with new malignancy between 1-10 weeks prior
* Are scheduled to receive cancer-directed therapy at Seattle Children's Hospital
* Has provided written informed consent (child aged 18 years and older), written assent (child aged 13-17 years), verbal assent (child aged 7-12 years).
* Able to speak and read English language
* Cognitively able to participate in interactive interviews

Exclusion Criteria:

* Parent is < 18 years of age
* Parent is cognitively or physically unable to participate in interactive interview
* Parent is unable to speak and read English language
* Parent or child participated on prior PRISM intervention study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Parent-Reported Resilience | 3 months

SECONDARY OUTCOMES:
Parent-reported Stress Survey Response | 3 months
Parent-reported psychological distress Survey Response | 3 months
Parent-reported social support Survey Response | 3 months
Parent-reported quality of life Survey Response | 3 months
Parent-reported benefit finding Survey Response | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rosenberg AR, Zhou C, Bradford MC, Barton K, Junkins CC, Taylor M, Kross EK, Curtis JR, Dionne-Odom JN, Yi-Frazier JP. Parent Perspectives after the PRISM-P Randomized Trial: A Mixed-Methods Analysis. J Palliat Med. 2021 Sep;24(10):1505-1515. doi: 10.1089/jpm.2020.0720. Epub 2021 Mar 15. PMID 33720787
- [Derived] Rosenberg AR, Bradford MC, Junkins CC, Taylor M, Zhou C, Sherr N, Kross E, Curtis JR, Yi-Frazier JP. Effect of the Promoting Resilience in Stress Management Intervention for Parents of Children With Cancer (PRISM-P): A Randomized Clinical Trial. JAMA Netw Open. 2019 Sep 4;2(9):e1911578. doi: 10.1001/jamanetworkopen.2019.11578. PMID 31532518